CLINICAL TRIAL: NCT02555514
Title: Identification of Biochemical and Biomechanical Markers for Cartilage Degeneration in the Knee Joint (IBBM-CKJ)
Acronym: IBBM-CKJ
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Dr. Jan Siewe (Other)
Responsible Party: Sponsor-Investigator, Dr. Jan Siewe, Dr.med., University of Cologne
Organization: University of Cologne (Other)
Other Study IDs: IBBM-CKJ
Record Dates: First submitted 2015-09-15; First posted 2015-09-21 (Estimated); Last update posted 2015-09-21 (Estimated); Status verified 2015-09

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — In order to investigate cartilage degeneration/turnover (COMP, collagen II, GAGs), miRNA and cytokine profiles 4 blood draws will be carried out
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Knee Osteoarthritis: The study population consists of 100 enrolled patients with different stages of knee OA and varus malalignment >4° with respect to the mechanical loading axis of the lower extremity. A minimum of 40 patients are to be included per year, so that the study period will be planned from January 1st, 2015 to June 30th, 2017. Preliminary results will be reviewed by the end of every year and intermediate reports will be generated by the sub-study-groups

SUMMARY:
The association between varus malalignment and dynamic knee loading / adduction moment and progression of knee joint cartilage degeneration in the lateral compartment is unclear and has not been studied in detail before. There is a need to identify relevant parameters explaining this cause-effect relationship. It is the purpose of the study to correlate load changes in knee joints with biomechanical and biochemical alterations in cartilage to understand the underlying mechanism of load induced cartilage degeneration in patients. This study will therefore include patients with different stages of knee OA with various malalignments. Moreover, analyzing changes in cartilage morphology, radiography and MRI and correlate those findings with alterations in biochemical parameters in cartilage, serum, urine and synovial fluid will allow us to identify novel biomarkers for the onset and progression of joint cartilage degeneration in varus malaligned knees.

The following hypotheses will be tested:

1. Knee joint cartilage degeneration progresses from medial to lateral in varus-aligned knees.
2. External knee adduction moments in patients with isolated medial OA are higher when compared with patients with OA of the medial and lateral compartment.
3. Morphological and mechanical properties of cartilage show different stages of degeneration when comparing the mechanically stronger loaded medial with the lateral compartment of the knee.
4. Histological and biochemical analysis of the cartilage indicate different stages of degeneration when comparing the mechanically loaded medial with the lesser loaded lateral compartment of the knee.
5. Synovial fluid analysis, as well as serum biomarkers of cartilage metabolism demonstrate cartilage degeneration and are related to biomechanical determinants of OA in the knee.
6. Novel biomarkers (ECM, miRNA, cytokines, mitochondria related, mechanical determinants) for varus-aligned knees can be identified.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a painful and debilitating disease of the synovial joints, affecting the structural and functional integrity of articular cartilage, subchondral bone, synovium and the adjacent supporting connective tissue . It is a degenerative disorder characterized by cartilage loss with high prevalence in individuals over an age of 55 years. The most affected region in OA is the medial compartment of the knee. The symptoms of OA include joint pain, stiffness, and swelling which may lead to impaired physical function and muscle weakness . The etiology of the disease is multifactorial and not fully understood. Traditionally, OA was regarded as a "wear and tear" disease caused by ageing, but both non-physiological mechanical loading (e.g. malalignment, obesity, trauma or joint instability) of a normal joint or physiological mechanical loading of a pathological joint can induce OA .

Joint misalignment has been identified as a potential biomechanical risk factor for development and progression of knee OA. Although determination of malalignment might provide important information about the load distribution in static conditions , dynamic loading parameters have been analyzed during gait to provide information about the total extrinsic load at the knee during the stance phase. According to Andriacchi, the external knee adduction moment can be used to predict load distribution between the medial and lateral compartments of the knee during dynamic activities. Increased external adduction moments are associated with increased joint forces on the medial plateau. During walking, forces are not evenly distributed across the joint surface and approximately 70% of the total load passes through the medial compartment. This may contribute to the higher prevalence of OA in this compartment . It can be expected that in patients with a varus deformity an even higher proportion of load is supported by the medial compartment. This may result in acceleration of articular cartilage degeneration.

The link between mechanical loading and the severity and progression of medial OA has been shown by many studies. Disease severity was found to correlate with the knee adduction moment , knee adduction angular impulse and knee extension moment . Miyazaki et al. analyzed the disease progression of OA patients during seven years. Patients that showed radiographic disease progression in the medial knee compartment also presented more severe knee pain and greater knee adduction moment than patients without disease progression. Baliunas et al. observed a significant greater knee adduction moment in OA patients with different levels of disease severity, but no significant differences were found in the sagittal moments. Thorp et al. analyzed not only the knee adduction moment but also the knee adduction angular impulse for the stance phase in healthy subjects and OA patients with mild and moderate disease progression in the medial knee compartment. The peak knee adduction moment and the knee adduction angular impulse were significant different between the control group, mild and moderate OA patients. Furthermore, the parameter knee adduction angular impulse was significantly different between mild and moderate OA patients, suggesting that this parameter can describe functional changes between different stages of disease progression.

While the relationship of varus malalignment and OA of the medial compartment is well described in the literature, little information is available if and how varus malalignment affects the lateral compartment. Fantini Pagani recently demonstrated that cartilage mechanical quality is not related to the knee adduction moment during gait in patients with severe OA.

Authors further reported that mechanical properties of osteoarthritic cartilage are highly variable indicating a complex relationship between joint loading and tissue changes during degenerative processes of articular cartilage. In clinical practice, patients with an identical mechanical varus malalignement of the lower extremity may show either isolated osteoarthritis of the medial compartment of the knee (example 1), or OA of the medial, lateral and patellofemoral compartment (example 2). This entity suggests that osteoarthritic disease in varus malaligned knees, in which the medial compartment is submitted to excessive overload, progress from medial to lateral over time. It could be assumed that mechanobiological factors and inflammatory reactions rather than mechanical load transmission play a major role in disease progression in the osteoarthritic knee.

Mechanobiological factors are thought to cause changes in articular cartilage thickness distributions in a joint throughout life . Healthy articular cartilage tends to be thickest in joints that experience high forces such as the knee. In addition, side differences in muscle cross sectional area positively correlated with side differences in articular cartilage morphology . Previous studies showed, that for healthy knees, the ratio of medial to lateral cartilage is greater in individuals that have a larger peak knee adduction moment during walking, suggesting that cartilage is thicker in areas where load is greater. These results are supported by those from animal studies in which articular cartilage increased in thickness by up to 19 to 23% when high mechanical loads were applied. An increase in cartilage thickness with exposure to higher loads may be off-set by a greater cartilage surface that may be caused by high physical activity during growth . Changes in tibio-femoral cartilage thickness are not dose-dependent suggesting that adult human cartilage morphology may not be sensitive to or improve with training .

Previous studies on animals and humans have shown that disuse like immobilization or strenuous mechanical loading induces changes in cartilage morphology and biology.

Cartilage composition and morphology is optimized for load-bearing function and characterized by the ability to sustain high and repetitive mechanical loads occurring during daily living. This mechanical function of cartilage is directly linked to the composition of the extracellular matrix (ECM). The synthesis and degradation of ECM molecules affect the mechanical properties of articular cartilage. The main ECM components are collagen II and non-collagenous proteins such as the proteoglycan aggrecan and other glycoproteins. Potential biological markers for cartilage metabolism include these matrix components and/or their breakdown products, cytokines, and proteases (eg. metalloproteases) and they can be quantified in serum, urine and synovial samples. Several serum biomarkers have been identified to monitor cartilage metabolism . One established biomarker for monitoring cartilage metabolism in relation to joint degeneration in OA , rheumatoid arthritis (RA) and injured knees is cartilage oligomeric matrix protein (COMP). In addition, previous studies have reported an increase in serum COMP concentration immediately after exercise with the dose of mechanical loads determining the magnitude and duration of increased serum COMP concentration. Besides COMP, biomarker of collagen II and aggrecan synthesis and degradation are suitable to monitor cartilage metabolism. Moreover, microRNAs can play a pivotal role for extracellular matrix homeostasis and are detectable at specific stages during OA progression. So far, miR-140, miR-9, miR-98 and miR-146 were found to be upregulated in osteoarthritic patient material and their expression is linked to the IL-1 beta induced production of TNF-alpha and matrix degradation in osteoarthritic cartilage . miRNAs can be released to the serum in various diseases and may have prognostic potential to determine the onset and progression of cartilage degeneration during OA. Finally, mitochondria damage is linked to reduced ECM production, secretion and enhanced degradation in cartilage. Recent reports show that specific inhibitors of the mitochondrial respiratory chain can suppress the synthesis of the ECM in articular chondrocytes and induced the production of proinflammatory cytokines and multiple factors released from damaged mitochondria, e.g damage mitochondrial DNA, reactive oxygen species, cytochrome c, proline/hydroxyproline synthesis, ATP and lactate production, could act as biomarkers for OA.

Inflammation within the joint of the knee is important in the pathophysiologic processes occurring after the onset of OA by high mechanical load. Cytokines are key players in the inflammatory mechanism and contribute to the progression of the cartilage damage. Therefore, the investigators focus on the effects of inflammation in OA and the role of pro-inflammatory and anti-inflammatory cytokines which can cause a deleterious or beneficial outcome. Investigation of the underlying mechanisms will help the investigators in understanding how cytokines contribute to the progression of OA and provide potential targets for novel therapeutics and biomarkers for diagnosis and prognosis of OA. Differences in the cytokine profile were reported for patients with OA, RA and healthy controls. Specific cytokines which are involved in OA were previously detected in blood as well as in synovial fluid . Cytokine expression in fluids may represent reliable diagnostic marker for early and late stages of OA. Recent data indicate potential correlations in the cytokine profile between blood and synovial fluid , which should be validated in the investigations. In addition, the investigators want to analyze the cytokine profile in tissue samples of OA and correlate the results with the profiles of serum and synovial fluid and clinical parameters. These results could link inflammatory reactions induced by the OA of the medial compartment to malalignment and to a progression of OA in the unaffected areas of the lateral compartments.

In summary, greater knee adduction moment is associated with greater load transmission through the medial knee compartment. Numerous studies identified increased knee adduction moment in patients with medial knee OA and varus deformity compared to healthy subjects. However, it is unclear how varus malalignment and dynamic knee loading / adduction moment affects the cartilage of lateral compartment. Morphological and biochemical markers are able to analyse cartilage degeneration in vivo in humans in relation to mechanical loading, a potential biomechanical risk factor for development and progression of knee OA.

ELIGIBILITY:
Inclusion Criteria:

* End stage medial, bi- or tricompartimental OA with indication to total knee replacement with failure of conservative treatment
* No more than mild symptoms of other joints in the lower limbs (VAS≤ 4)
* Age > 18 years
* BMI < 35

Written informed consent must be obtained from all patients prior to any study-related procedure.

Exclusion Criteria:

* BMI ≥ 35
* Post-infectious condition of the affected knee
* Valgus- or neutral lower limb axis
* Pacemaker or any other medical condition that does not allow MRI scans
* Systemic arthritic conditions
* Previous surgery of lower extremities and/or low back within the last 6 months
* Musculoskeletal or neurological condition severely affecting lower limb function
* Contraindications to MRI
* Not able to walk independently without a walking aid
* Additional infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: End stage medial, bi- or tricompartimental OA with indication to total knee replacement with failure of conservative treatment
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
measurement of Knee joint cartilage degeneration progresses from medial to lateral in varus-aligned knees in mm . | Change from Baseline 12 month
  The association between varus malalignment and dynamic knee loading / adduction moment and progression of knee joint cartilage degeneration in the lateral compartment is unclear and has not been studied in detail before. There is a need to identify relevant parameters explaining this cause-effect relationship. It is the purpose of the study to correlate load changes in knee joints with biomechanical and biochemical alterations in cartilage to understand the underlying mechanism of load induced cartilage degeneration in patients. This study will therefore include patients with different stages of knee OA with various malalignments. Moreover, analyzing changes in cartilage morphology, radiography and MRI and correlate those findings with alterations in biochemical parameters in cartilage, serum, urine and synovial fluid will allow us to identify novel biomarkers for the onset and progression of joint cartilage degeneration in varus malaligned knees.